CLINICAL TRIAL: NCT07285486
Title: Regenerative Peripheral Nerve Interfaces for the Treatment of Painful Neuromas in Major Limb Amputees
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Theodore Alexander Kung, Principal Investogator, University of Michigan
Other Study IDs: HUM00120915
Record Dates: First submitted 2025-12-02; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Amputation Neuroma
MeSH Terms: interventions — Amputation, Surgical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Amputation Pain: Participants who were existing amputees who had chronic neuroma pain at the amputation site.
  Interventions: Procedure: Amputation with Regenerative Peripheral Nerve Interfaces (RPNI)
- Prophylactic Treatment Group: Participants who had a lower extremity amputated during the study and were prophylactically treated for pain.
  Interventions: Procedure: Amputation with Regenerative Peripheral Nerve Interfaces (RPNI); Other: Amputation Without RPNI

INTERVENTIONS:
Procedure: Amputation with Regenerative Peripheral Nerve Interfaces (RPNI) — Free-muscle graft over cut nerve ends for treatment of neuromas at site of an amputation.
  Other Names: RPNI
Other: Amputation Without RPNI — Standard of care for lower-extremity amputation
  Groups: Prophylactic Treatment Group

SUMMARY:
The Regenerative Peripheral Nerve Interface (RPNI) is a novel strategy to prevent neuroma formation in transected peripheral nerves. The RPNI consists of a residual peripheral nerve that is implanted into a free skeletal muscle graft either at the time of limb amputation or after excision of a terminal neuroma bulb. The sprouting axons of the nerve readily reinnervate the free muscle graft, thereby greatly reducing the chance of neuroma formation.

This investigation has a prospective cohort study design involving major lower limb amputees drawn from both the University of Michigan Health Systems and VA Health System of Ann Arbor. To objectively evaluate the effect of RPNI surgery on patients' perception of pain and to measure other health-related quality of life metrics relating to neuroma pain, this clinical trial will utilize specific, validated patient-reported outcomes measures (PROMs) to assess targeted domains in patients with major limb amputation. These survey instruments will determine: 1) patterns of pain medication use, including the use of opioids, 2) functional status and use of a prosthetic device, 3) changes in neuroma pain quality, 4) limitations in activities of daily living due to neuroma pain, 5) depression and anxiety relating to neuroma pain.

ELIGIBILITY:
Inclusion Criteria:

* Major lower limb amputation (chronic pain treatment group only)
* Symptomatic residual limb neuroma (chronic pain treatment group only)
* Undergoing a major lower limb amputation (prophylactic pain treatment group only)

Exclusion Criteria:

* History of chronic amputation-related pain (prophylactic pain treatment group only)
* History of regenerative peripheral nerve interface (RPNI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants were recruited from plastic surgery, orthopedic surgery, and vascular surgery clinics.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Orthotics and Prosthetics Users Survey (OPUS) | Up to 12 months postoperatively
  The OPUS was a self-report questionnaire consisting of five modules. It can be used for prosthetic and orthotic programs for quality assessment, to maintain awareness of improvement in activities, to evaluate changes in patient's functional status and quality of life, and to assess satisfaction with devices and services. This study used the Functional Status Measure module, which was a 20-question survey that used a Likert scale ranging from 1 (very easy) to 5 (cannot do this activity).
Pain Cognition Scale (PCS) | Up to 12 months postoperatively
  The PCS evaluated the relationship between thoughts and pain. The PCS was a 13-question survey that used a Likert scale ranging from 0 (not at all) to 4 (all the time). Total score ranged from 0 (no pain catastrophizing) to 52 (highest level of pain catastrophizing), with a score of 30 indicating a clinically high level of pain catastrophizing.
Short-form McGill Pain Questionnaire 2 (SF-MPQ-2) | Up to 12 months postoperatively
  The SF-MPQ-2 was a pain assessment tool that measured both neuropathic and non-neuropathic pain. It used 22 descriptors, grouped into four subscales (continuous, intermittent, neuropathic, and affective) along with a Present Pain Intensity (PPI) scale. The descriptors and PPI all used a Likert scale that ranged from 0 (none) to 10 (worst possible). The SF-MPQ-2 was scored by calculating the average ratings for each of the four subscales and the total pain score and averaging all 22 item ratings, resulting in a score ranging from 0 (none) to 10 (worst possible).
Patient-Reported Outcomes Measurement Information System (PROMIS) - Pain Interference | Up to 12 months postoperatively
  The PROMIS was a system of standardized, scientifically validated questions used to measure a patient's physical, mental, and social health status. The PROMIS pain interference short form had 6 questions ranging from 1 [not at all] to 5 [very much]. The PROMIS was scored by summing the values of the responses within each short form. The raw score was converted to a standardized T-score using specific scoring tables found in the instrument's scoring manual.
PROMIS - Neuropathic Pain Quality | Up to 12 months postoperatively
  The PROMIS was a system of standardized, scientifically validated questions used to measure a patient's physical, mental, and social health status. The PROMIS neuropathic pain quality short form had 5 questions ranging from 1 [not at all] to 5 [very much]. The PROMIS was scored by summing the values of the responses within each short form. The raw score was converted to a standardized T-score using specific scoring tables found in the instrument's scoring manual.
PROMIS Pain Intensity | Up to 12 months postoperatively
  The PROMIS was a system of standardized, scientifically validated questions used to measure a patient's physical, mental, and social health status. The PROMIS pain intensity short form had 3 questions ranging from 0 [had no pain] to 5 [very severe]. The PROMIS was scored by summing the values of the responses within each short form. The raw score was converted to a standardized T-score using specific scoring tables found in the instrument's scoring manual.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) - Depression | Up to 12 months postoperatively
  The PHQ-9 was a nine-question self-report questionnaire used to screen for depression, diagnose its severity, and monitor treatment response. Each of the nine questions was scored on a four-point scale from 0 ("Not at all") to 3 ("Nearly every day"). The PHQ-9 asked about the frequency of specific depressive symptoms over the past two weeks, with a total score ranging from 0 to 27, with scores below 5 indicating no depression and scores above 20 indicating severe depression.
General Anxiety Disorder-7 (GAD-7) - anxiety | Up to 12 months postoperatively
  The GAD-7 was a seven-item questionnaire used to screen for and measure the severity of generalized anxiety disorder (GAD). It asked about symptoms like feeling nervous, worrying too much, and trouble relaxing, with responses scored from 0 to 3 for each of the seven questions. The total score, ranging from 0 to 21, is interpreted to indicate the level of anxiety: 0-4 (minimal), 5-9 (mild), 10-14 (moderate), and 15-21 (severe).
Fibromyalgia Survey Questionnaire (FSQ) | Up to 12 months postoperatively
  The FSQ was a tool used to assess the key symptoms of fibromyalgia by evaluating widespread pain and the severity of other somatic symptoms. It was comprised of two tools, the widespread pain index (WPI) subsection and the symptom severity score (SSS), which were summed to get a result. The WPI asked participants to mark off from a list of 19 potential pain locations on a body diagram. which were summed. The total score ranged from 0 to 19. The SSS evaluated the severity of three major symptoms and the severity of other somatic symptoms. The SSS consisted of 6 questions with a total score ranging from 0 to 12. The total range of both tools combined was 0 to 31, with a total score of ≥13 supporting a diagnosis of fibromyalgia.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Kung, MD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Department of Veterans Affairs Ann Arbor Health System, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee JC, Kubiak CA, Best CSW, Hamill JB, Ki J, Kim HM, Roth RS, Kozlow JH, Tinney MJ, Geisser ME, Cederna PS, Kemp SWP, Kung TA. Regenerative Peripheral Nerve Interface Surgery to Treat Chronic Postamputation Pain: A Prospective Study in Major Lower Limb Amputation Patients. Ann Surg Open. 2025 Jan 7;6(1):e535. doi: 10.1097/AS9.0000000000000535. eCollection 2025 Mar. PMID 40134500